CLINICAL TRIAL: NCT05796908
Title: A Prospective, Multi-Center, Single-Arm Clinical Trial of the Safety and Effectiveness of the Aptis PRUJ Prosthesis for the Treatment of Patients With Proximal Radial Ulna Joint Disorders.
Brief Title: Aptis PRUJ Prosthesis for the Treatment of Patients With Proximal Radial Ulna Joint Disorders.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aptis Medical (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AP-PRO-001
Record Dates: First submitted 2023-03-10; First posted 2023-04-04 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Arthritis; Unstable Radial Head; Proximal Radioulnar Joint Instability; Decreased Motion at the Proximal Radioulnar Joint and/or the Radio-humeral Joint
Keywords: PRUJ; Disorders; radio-humeral joint; proximal radioulnar joint
MeSH Terms: conditions — Arthritis; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Aptis PRUJ Prothesis (Experimental): Investigational Aptis PRUJ Prothesis treatment
  Interventions: Device: Aptis PRUJ Prosthesis

INTERVENTIONS:
Device: Aptis PRUJ Prosthesis — A prosthetic implant for replacement of the proximal radial ulna joint.

SUMMARY:
A Prospective, Multi-Center, Single-Arm Clinical Trial of the safety and effectiveness of the Aptis PRUJ prosthesis for the treatment of patients with proximal radial ulna joint disorders

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm clinical trial of the safety and effectiveness of the Aptis PRUJ prosthesis for the treatment of patients with proximal radial ulna joint disorders. A total of 84 patients will be enrolled in this trial with 9 centers participating in the US. The total study duration will be approximately 36 months, with an enrollment period of 12 months, followed by a 24 month follow-up period. Annual visits will continue until the last patient reaches the 2-year post-operative time point.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, subjects must meet all of the following criteria:

  1. Patient is skeletally mature and under 85 years of age.
  2. Patient has a painful, unstable radial head due to degeneration or post-traumatic disabilities presenting pain, crepitation, and decreased motion at the radiohumeral and/or proximal radioulnar joint and is otherwise
  3. Patients willing and able to understand and sign the informed consent. In the opinion of the Investigator, the patient has the understanding and willingness to comply with all study requirements including the post-operative rehabilitation and follow-up visits per protocol.

Exclusion Criteria:

* 1. Inadequate bone stock or soft tissue coverage 2. Patients with severe humeral/ulnar arthritis, defined as:

  1. Pain at terminal flexion/extension
  2. Pain throughout ROM with loss of motion in terminal flexion and/or extension 3. Patients with an allergy to the implant materials 4. Active systemic infection or infection at the site of surgery 5. Physical interference with or by other prostheses during implantation or use 6. Have a Body Mass Index (BMI) greater than 35 kg/m2 7. Have any mental or psychological disorder that would impair the ability to complete the study questionnaires 8. Have significant comorbidities or conditions associated with high-risk for surgical or anesthetic survival (e.g., renal failure, peripheral vascular disease, unstable cardiac disease, poorly controlled diabetes, immunosuppression, etc.) 9. Have any medical condition or other circumstances that might interfere with the ability to return for follow-up visits in the judgment of the Investigator, including any systemic illness, neuromuscular, neurosensory, or musculoskeletal deficiency that would render the subject unable to perform appropriate post-operative rehabilitation 10. Have any condition which, in the judgment of the Investigator, would preclude adequate evaluation of the device's safety and performance 11. Skin, bone, circulatory and/or neurological deficiency at or affecting the implantation site 12. Prisoners 13. Patients on chronic corticosteroid or non-steroidal anti-inflammatory therapy 14. Women who are pregnant or breast-feeding or are planning to become pregnant during the study.

     15. Patients with a documented history of uncontrolled diabetes. 16. Patients with known allergies against anesthesia. 17. Patients with a history of or current drug and/or alcohol abuse 18. Patients unlikely to cooperate or are legally incompetent. 19. Patients with legal involvement, including an active claim for workman's compensation, or any other issue that would hinder completion of the two-year follow period.

     20. Patients who are participating or have participated in any other study involving an investigational drug or device within the past 3 months.

     Intra-operative Exclusion Criteria

     Subjects who meet any of the following intra-operative screening criteria will be excluded from participation in this study:
     * A proximal radio ulnar joint that cannot be reduced intraoperatively
     * Inadequate bone quality that would allow for implant placement
     * Not enough radius bone proximally for device implantation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Sucess | 24 months
  A non-inferiority composite primary endpoint for effectiveness and safety, where a subject is considered a success if they meet the following criteria:
  * Mayo Elbow Performance Score, where success is defined as Good or Excellent at 24 months; and
  * Absence of radiographic evidence of periprosthetic osteolysis (radiolucent line >2mm around entire radial stem and ulnar screws), and no screw breakage at 24 months; and
  * Absence of device-related serious adverse events including any revisions and removals through 24 months

SECONDARY OUTCOMES:
Effectiveness | 6 weeks, 3 months, 6 months, 12 months, 24 months
  The following secondary endpoints will evaluate the effectiveness of the investigational device:
  * Pre- vs. Post-operative function assessed via Mayo Elbow Performance Score
  * Mayo Subscores
    * Pain
    * Range of motion
    * Instability
    * Function
Effectiveness | 6 weeks, 3 months, 6 months, 12 months, 24 months
  Changes in overall health at all follow-up time points assessed via SF-36
Effectiveness | 6 weeks, 3 months, 6 months, 12 months, 24 months
  Change in disability index assessed at all follow-up time points via DASH
Radiographic | 6 weeks, 3 months, 6 months, 12 months, 24 months
  Radiolucencies around radial stem and ulnar screws
Radiographic | 6 weeks, 3 months, 6 months, 12 months, 24 months
  Subsidence of radial component
Radiographic | 6 weeks, 3 months, 6 months, 12 months, 24 months
  Screw breakage
Radiographic | 6 weeks, 3 months, 6 months, 12 months, 24 months
  Ulnar variance
Health Economic | 6 weeks, 3 months, 6 months, 12 months, 24 months
  Use of other concomitant medications
Health Economic | 6 weeks, 3 months, 6 months, 12 months, 24 months
  Post-operative recovery time (return to daily activities/work)
Health Economic | 6 weeks, 3 months, 6 months, 12 months, 24 months
  Post-operative rehabilitation details

CONTACTS AND LOCATIONS:
Overall Officials: John Scheker, Study Chair — Aptis Medical
Locations (6):
- United States (6):
  - Indiana Hand to Shoulder Center, Carmel, Indiana
  - Kleinert Kutz Hand Care Center, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Orthopedic Associates of Southwest Ohio, Dayton, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No